CLINICAL TRIAL: NCT05636839
Title: UVB-induced Treg Cells Exert Antigen-specific Suppression Through LAG-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202112019RINA
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2021-12

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: UVB treatment; antigen specificity; regulatory T cell; mass cytometry
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UVB treatment (Experimental): UVB treatment 3 times per week for 10 weeks
  Before treatment starts, researchers will collect 20 ml of blood from participants. After 10-week treatment, researchers will collect 20 ml of blood from participants again.
  Interventions: Radiation: UVB treatment

INTERVENTIONS:
Radiation: UVB treatment — UVB treatment 3 times per week for 10 weeks

SUMMARY:
The goal of this clinical trial is to compare the immune cell population in blood of the participants with psoriasis/atopic dermatitis before and after UVB treatment. The main questions it aims to answer are:

1. how immune cells in the PBMCs from blood of participants are affected by UVB treatment
2. will UVB treatment expand the antigen-specific Treg cell population
3. will UVB treatment enhance the suppressive function of Treg cells

Participants giving written informed consent will donate their blood (20 ml) before UVB treatment begins. After 8 to 10-week treatment course, the participants will donate their blood (20 ml) again.

Researchers will compare immune cell population changes in the PBMCs of participants before and after UVB treatment. In addition, researchers will purify Treg cells from participant blood before and after UVB treatment to test their suppressive activity by ex vivo suppression assay.

DETAILED DESCRIPTION:
UVB irradiation suppresses immune responses partly via the induction of Treg cells. However, it is still not clear whether the therapeutic effect of UVB to treat skin inflammatory diseases (such as psoriasis and atopic dermatitis) results from the increase of Treg cell population. In addition, how UVB induces antigen-specific Treg cells needs to be elucidated.

In this study, researchers will examine the Treg cell population in the blood of participants with psoriasis or atopic dermatitis under UVB treatment. We will analyse changes of immune cell populations in the blood of participants using mess cytometry. We will also investigate the suppressive function of Treg cells sorted from peripheral blood mononuclear cells (PBMCs) to see whether UVB treatment will affect the function of Treg cells.

Enrolled participants will donate 20 ml of blood before UVB treatment begins. They will receive UVB irradiation 2 to 3 times per week, and the treatment course will last 8 to 10 weeks, which is defined as a complete treatment. After a complete treatment, the participants will donate 20 ml of blood again, and the trial ends.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age
2. Able and willing to provide written informed consent

Exclusion Criteria:

1. UV exposure in the last 8 weeks before study entry
2. Patients with contraindications for UV-treatment
3. History of cancer and primary immunodeficiency
4. pregnant or nursing mother
5. participating in another clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of Treg cells | 10 weeks
  Change from baseline in Treg cell percentage in the peripheral blood of psoriasis patients treated with UVB

CONTACTS AND LOCATIONS:
Overall Officials: Yungling Lee, Dr, Principal Investigator — Academia Sinica, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No